CLINICAL TRIAL: NCT03626740
Title: Experimental Research on Deep Carious Lesion Treatment of Permanent Molars in Children, Aiming to Preserve Dental Pulp Vitality
Brief Title: Experimental Research on Deep Carious Lesion Treatment of Molars
Acronym: VITAPULP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Andreea Didilescu, DDS, Vice dean for Research, Professor, Carol Davila University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PN-III-P4-ID-PCE-2016-0506
Record Dates: First submitted 2018-08-01; First posted 2018-08-13 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Dental Caries in Children
Keywords: dental pulp; deep carious lesions; treatment effect
MeSH Terms: interventions — TheraCal; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TheraCal (Experimental): Indirect pulp capping with TheraCal
  Interventions: Other: TheraCal
- Mineral trioxide aggregate (MTA) (Active Comparator): Indirect pulp capping with MTA
  Interventions: Other: MTA

INTERVENTIONS:
Other: TheraCal — Caries removal without pulp exposure (stepwise excavation) followed by indirect pulp capping with TheraCal
  Arms: TheraCal
Other: MTA — Caries removal without pulp exposure (stepwise excavation) followed by indirect pulp capping with MTA
  Arms: Mineral trioxide aggregate (MTA)

SUMMARY:
Maintaining dental pulp vitality is crucial for tooth preservation and functionality. Untreated dental caries may lead to pulp necrosis and infection, affecting children's growth and well-being. The first permanent teeth erupt around 6 years old. These are the first molars (FPM), which are frequently affected by caries, soon after their eruption.

In the present application, our main goal is to determine whether two treatment groups (MTA and TheraCal) are long-term effective in preserving pulp vitality among children' FPM affected by deep caries.

DETAILED DESCRIPTION:
Among the most frequently used materials for pulp capping are calcium hydroxide, mineral trioxide aggregate (MTA), and, more recent, TheraCal. All of them are biocompatible and induce the formation of coronal hard tissue barriers (tertiary reparative dentin). Calcium hydroxide, considered for a long time the gold standard of direct pulp capping materials, has excellent antibacterial and remineralisant properties; however, it lacks adhesion, especially at moist dentin, and reparative dentin is less homogenous.

MTA proved to stimulate protective dentin bridge formation without inflammatory changes and least necrosis. It is also moisture tolerant, but it is more expensive, has poor handling characteristics and slow setting time.

TheraCal bonds to deep moist dentin, has strong physical properties, no solubility, high radioopacity and higher calcium releasing abilities than MTA or calcium hydroxide.

ELIGIBILITY:
Inclusion Criteria:

* untreated deep uncomplicated carious lesions in first permanent molars (FPM)
* absence of clinical diagnosis of pulp exposure
* fistula
* swelling of periodontal tissues
* abnormal tooth mobility
* history of spontaneous pain or sensitivity to percussion
* healthy appearance of adjacent gingiva
* normal tooth color
* positive vitality to thermal and electric tests.

Exclusion Criteria:

* FPM with previous treatment
* FPM with developmental abnormalities (such as enamel hypoplasia, dentinogenesis imperfecta etc.)
* children with mental disabilities or systemic diseases.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-04 (Actual)

PRIMARY OUTCOMES:
Clinical pulpal survival rate | 20 months
  Pulpal survival is defined by positive response without lingering sensation to the cold test, absence of clinical signs and symptoms, and no apical radiolucency on the periapical radiograph.

SECONDARY OUTCOMES:
Incidence of apical root maturation (apexogenesis) | 20 months
  We will investigate the treatment effect on apexogenesis in children who had incomplete root formation at the beginning of the study and preserve their pulp vitality at the end of the study. The outcome will be compared radiographically with apical maturation in molar pairs (healthy contralateral molar, where applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Andreea C Didilescu, DDS, PhD, Principal Investigator — Carol Davila University of Medicine and Pharmacy
Locations (1):
- Division of Pedodontics, Faculty of Dental Medicine, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No